CLINICAL TRIAL: NCT01864902
Title: Clinical Study of Chimeric CD(Cluster of Differentiation)33 Antigen Receptor-modified T Cells in Relapsed and/or Chemotherapy Refractory Acute Myeloid Leukemias
Brief Title: Treatment of Relapsed and/or Chemotherapy Refractory CD33 Positive Acute Myeloid Leukemia by CART-33
Acronym: CART33
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, PI, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-006
Record Dates: First submitted 2013-05-20; First posted 2013-05-30 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Relapsed Adult Myeloid Leukemia; Chemotherapy Refractory Adult Myeloid Leukemia
Keywords: CD33 positive acute myeloid leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid | interventions — Immunotherapy, Adoptive; Sensitivity and Specificity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-CD33 CAR T cells (Experimental): Patients receive anti-CD33-CAR retroviral vector-transduced autologous or donor-derived T cells on days 0,1, 2 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: CART33 cells; Biological: anti-CD33 CART; Biological: anti-CD33 CAR T cells

INTERVENTIONS:
Biological: CART33 cells — genetically modified lymphocyte therapy
  Other Names: chimeric antigen receptor T cells with specificity for CD33
Biological: anti-CD33 CART
  Other Names: CART33
Biological: anti-CD33 CAR T cells

SUMMARY:
RATIONALE: Placing a tumor antigen chimeric receptor that has been created in the laboratory into patient autologous or donor-derived T cells may make the body build immune response to kill cancer cells.

PURPOSE: This clinical trial is to study genetically engineered lymphocyte therapy in treating patients with CD33 positive acute myeloid leukemias that is relapsed (after stem cell transplantation or intensive chemotherapy) or refractory to further chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and feasibility of the chimeric antigen receptor T cells transduced with the anti-CD33 vector (referred to as CART-33 cells).

II. Determine duration of in vivo survival of CART-33 cells. RT-PCR (reverse transcription polymerase chain reaction) analysis of whole blood will be used to detect and quantify survival of CART-33 TCR zeta:CD137 and TCR (T-cell receptor) zeta cells over time.

SECONDARY OBJECTIVES:

I. For patients with detectable disease, measure anti-leukemia response due to CART-33 cell infusions.

II. To determine if the CD137 transgene is superior to the TCR zeta only transgene as measured by the relative engraftment levels of CART-33 TCR zeta:CD137 and TCR zeta cells over time.

III. Estimate relative trafficking of CART-33 cells in bone marrow.

IV. For patients with stored or accessible leukemia blasts, determine leukemia cell killing by CART-33 cells in vitro.

V. Determine if cellular or humoral host immunity develops against the murine anti-CD33, and assess correlation with loss of detectable CART-33 (loss of engraftment).

VI. Determine the relative subsets of CART-33 T cells (Tcm, Tem, and Treg).

OUTLINE: Patients are assigned to 1 group according to order of enrollment.

Patients receive anti-CD33-CAR (coupled with CD137 and CD3 zeta signalling domains)vector-transduced autologous T cells on days 0,1, and 2 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed intensively for 6 months, every 3 months for 2 years, and annually thereafter for 13 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with CD33+ acute myeloid leukemia in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled

  * CD33+ acute myeloid leukemia CR can not be achieved after at least 2 prior combination chemotherapy regimens.

AML in CR(complete remission)2 or CR3 and not eligible for allogeneic SCT because of age, comorbid disease, or lack of available family member or unrelated donor.

Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval < 1 year).

Relapsed after prior autologous or allogenic SCT. AML patients with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT.

Residual disease after primary therapy and not eligible for autologous SCT

* Expected survival > 12 weeks
* Creatinine < 2.5 mg/dl
* ALT(alanine aminotransferase)/AST (aspartate aminotransferase)< 3x normal
* Bilirubin < 2.0 mg/dl
* Any relapse after prior SCT will make patient eligible regardless of other prior therapy
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women

  * The safety of this therapy on unborn children is not known
  * Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
  * Uncontrolled active infection
  * Active hepatitis B or hepatitis C infection
  * Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
  * Previously treatment with any gene therapy products
  * Feasibility assessment during screening demonstrates < 30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD137 costimulation
  * Any uncontrolled active medical disorder that would preclude participation as outlined
  * HIV infection

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | Until week 24
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
Anti-leukemia responses to CART-33 cell infusions | up to 24 weeks

OTHER OUTCOMES:
in vivo existence of CART33 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Pediatrics Department of Chinese PLA General Hospital, Hematological Department, Affiliated Hospital of Changzhi Medical College, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang QS, Wang Y, Lv HY, Han QW, Fan H, Guo B, Wang LL, Han WD. Treatment of CD33-directed chimeric antigen receptor-modified T cells in one patient with relapsed and refractory acute myeloid leukemia. Mol Ther. 2015 Jan;23(1):184-91. doi: 10.1038/mt.2014.164. Epub 2014 Sep 1. PMID 25174587